CLINICAL TRIAL: NCT04132557
Title: Suicidality, Psychosis or Substance Abuse With Methylphenidate, Atomoxetine, Amphetamine/Dextroamphetamine or Lisdexamfetamine, a Post-authorization Safety Study
Brief Title: A Study on Suicidality, Psychosis or Substance Abuse With Methylphenidate, Atomoxetine, Amphetamine/Dextroamphetamine or Lisdexamfetamine
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108701; PCSESP002036 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Lisdexamfetamine Dimesylate; Atomoxetine Hydrochloride; Amphetamine; Dextroamphetamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Cohort 1 (Target): Methylphenidate Monotherapy: Participants will be analyzed for Attention Deficit Hyperactive Disorder (ADHD) who are new users of methylphenidate monotherapy. Analysis of data will be performed between 1 January 2001 to 30 September 2018.
  Interventions: Drug: Methylphenidate
- Cohort 2 (Comparator [C]): Lisdexamfetamine Monotherapy: Participants will be analyzed for ADHD who are new users of lisdexamfetamine monotherapy. Analysis of data will be performed between 1 January 2001 to 30 September 2018.
  Interventions: Drug: Lisdexamfetamine
- Cohort 3 (C): Atomoxetine Monotherapy: Participants will be analyzed for ADHD who are new users of atomoxetine monotherapy. Analysis of data will be performed between 1 January 2001 to 30 September 2018.
  Interventions: Drug: Atomoxetine
- Cohort 4 (C):Amphetamine/Dextroamphetamine Combo Therapy: Participants will be analyzed for ADHD who are new users of amphetamine/dextroamphetamine combo therapy. Analysis of data will be performed between 1 January 2001 to 30 September 2018.
  Interventions: Drug: Amphetamine; Drug: Dextroamphetamine

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate is common ADHD medications in the United States. This is a non-interventional study and no drug will be given as part of this study. Analysis will be performed from data taken from three United States (US) health care databases and one US electronic health record database.
  Groups: Cohort 1 (Target): Methylphenidate Monotherapy
Drug: Lisdexamfetamine — Lisdexamfetamine is common ADHD medications in the United States. This is a non-interventional study and no drug will be given as part of this study. Analysis will be performed from data taken from three US health care databases and one US electronic health record database.
  Groups: Cohort 2 (Comparator [C]): Lisdexamfetamine Monotherapy
Drug: Atomoxetine — Atomoxetine is common ADHD medications in the United States. This is a non-interventional study and no drug will be given as part of this study. Analysis will be performed from data taken from on three US health care databases and one US electronic health record database.
  Groups: Cohort 3 (C): Atomoxetine Monotherapy
Drug: Amphetamine — Amphetamine is common ADHD medications in the United States. This is a non-interventional study and no drug will be given as part of this study. Analysis will be performed from data taken from on three US health care databases and one US electronic health record database.
  Groups: Cohort 4 (C):Amphetamine/Dextroamphetamine Combo Therapy
Drug: Dextroamphetamine — Dextroamphetamine is common ADHD medications in the United States. This is a non-interventional study and no drug will be given as part of this study. Analysis will be performed from data taken from on three US health care databases and one US electronic health record database.
  Groups: Cohort 4 (C):Amphetamine/Dextroamphetamine Combo Therapy

SUMMARY:
The purpose of this study is to estimate the observed incidence of the health outcomes (suicide attempt or ideation, suicide ideation, suicide attempt, psychosis, and substance abuse) in a cohort of participants diagnosed with attention deficit hyperactivity disorder (ADHD) who are first-line new therapy with methylphenidate monotherapy, lisdexamfetamine monotherapy, atomoxetine monotherapy, amphetamine/dextroamphetamine combo therapy, and either methylphenidate/lisdexamfetamine/atomoxetine monotherapy or amphetamine/dextroamphetamine combo therapy during the 'on treatment' period from 7 days after the start of exposure through the end of exposure (treatment discontinuation for at least 60 days) and the 'intent to treat' period from 7 days after start of treatment to end of continuous observation; and to compare the hazards of outcomes (suicide attempt or ideation, suicide ideation, suicide attempt, psychosis, and substance abuse) in the target cohort (participants diagnosed with ADHD who are first-line monotherapy new users of methylphenidate) versus each comparator cohort (patients diagnosed with ADHD who are first-line newly exposed to lisdexamfetamine monotherapy, atomoxetine monotherapy, amphetamine/dextroamphetamine combo therapy) during the 'on treatment' period from 7 days after the start of exposure through the end of exposure (treatment discontinuation for at least 60 days) and the 'intent to treat' period from 7 days after start of treatment to end of continuous observation.

ELIGIBILITY:
Inclusion Criteria:

* New users of methylphenidate monotherapy or lisdexamfetamine monotherapy or atomoxetine monotherapy or amphetamine/dextroamphetamine combo therapy
* Prior diagnosis of ADHD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise of participants with attention deficit/hyperactivity disorder (ADHD) described in on three US health care databases and one US electronic health record which has data available through 1 January 2001 to 30 September 2018.
Sampling Method: Probability Sample
Enrollment: 430000 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Number of Incidence of Suicide Attempt or Ideation | Up to 17.8 years
  Number of incidence of suicide attempt or ideation will be reported. Analysis will be performed from data taken from three United States (US) health care databases and one US electronic health record database.
Number of Incidence of Suicide Attempt | Up to 17.8 years
  Number of incidence of suicide attempt will be reported. Analysis will be performed from data taken from three US health care databases and one US electronic health record database.
Number of Incidence of Suicide Ideation | Up to 17.8 years
  Number of incidence of suicide ideation will be reported. Analysis will be performed from data taken from three US health care databases and one US electronic health record database.
Number of Incidence of Psychosis diagnosis Followed by Anti-psychotic Drug Within 60 days | Up to 17.8 years
  Number of incidence of psychosis diagnosis followed by anti-psychotic drug within 60 days will be reported. Analysis will be performed from data taken from three US health care databases and one US electronic health record database.
Number of Incidence of Substance Abuse | Up to 17.8 years
  Number of incidence of substance abuse (excluding alcohol and nicotine) will be reported. Analysis will be performed from data taken from three US health care databases and one US electronic health record database.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Development, LLC Clinical Trial, Study Director — Janssen Research and Development LLC
Locations (1):
- Janssen Investigative Site, Titusville, New Jersey, United States